CLINICAL TRIAL: NCT03134716
Title: Role of Microglia in the Pathogenesis of Progressive Multiple Sclerosis
Acronym: PROMS
Status: Active, not recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: T99/2016
Record Dates: First submitted 2016-04-14; First posted 2017-05-01 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Correlation of blood biomarkers and MS progression
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Clinical follow-up: Clinical follow-up of MS-patients for 5 years. PET imaging data with PK11195 and TMSX only in baseline and with UCB-J at 5 years
- Healthy controls: comparison of healthy controls' and MS patients' PET imaging data with PK11195 and TMSX only in baseline and with UCB-J at 5 years

SUMMARY:
Our aim is to evaluate whether translocator binding protein (TSPO)-imaging correlates to Expanded Disability Status Scale (EDSS) and other disease progression-related clinical and paraclinical parameters in a homogenous cohort of 40-50-year old MS-patients, who are at risk of progression. The A2A-AR expression in this cohort will also be studied using the adenosine A2A-receptor (A2A-AR)-binding radioligand 11C-TMSX. The study cohort will also form the basis for a later follow-up study, which will be performed to evaluate the prognostic value of baseline TSPO-imaging in terms of disease progression. TSPO-imaging could thus be used as an imaging biomarker to help identifying patients to therapeutically prevent progression of MS. At the 5 year time point synaptic density will be evaluated using 11C-UCB-J radioligand and PET imaging.

DETAILED DESCRIPTION:
Protocol title: Role of microglia in the pathogenesis of progressive multiple sclerosis

Rationale of the study: The investigators have demonstrated earlier a statistically significant correlation between TSPO-binding and EDSS in a heterogeneous MS-population comprising both early RRMS and late secondary progressive multiple sclerosis (SPMS) patients. Now the investigators aim to evaluate whether TSPO-imaging correlates to EDSS and other disease progression-related clinical and paraclinical parameters in a homogenous cohort of 40-50-year old MS-patients, who are at risk of progression. The A2A-AR expression in this cohort will also be studied using the A2A-AR-binding radioligand 11C-TMSX. The study cohort will also form the basis for a later follow-up study, which will be performed to evaluate the prognostic value of baseline TSPO-imaging in terms of disease progression. TSPO-imaging could thus be used as an imaging biomarker to help identifying patients to therapeutically prevent progression of MS. At the 5 year time point synaptic density will be evaluated using 11C-UCB-J radioligand and PET imaging.

Study population: The study population will consist of a clinically homogenous group of 25 relapsing remitting multiple sclerosis (RRMS) patients with MS-diagnosis for at least 5 years, age 40-50 years, who may be using any first-line MS therapy. The patients will be recruited from the outpatient clinic of the Division of Clinical Neurosciences of the University Hospital of Turku, Finland. In addition the investigators will image a group of 10 age- and sex-matched healthy control subjects for comparison.

Study Objectives Primary: To evaluate how TSPO-ligand binding in the normal appearing white matter (NAWM) correlates to EDSS.

Secondary: 1) To evaluate how TSPO-ligand binding in the NAWM at baseline correlates to other standard clinical and paraclinical parameters typically associated with disease progression 2) To evaluate how 11C-TMSX-binding (to A2A-AR) correlates to the clinical and paraclinical parameters, and to TSPO-binding. 3) To evaluate how synaptic density evaluated using 11C-UCB-J binding correlates to patients cognitive functions.

Inclusion criteria: RRMS, age 40-50 years, MS-diagnosis for a minimum of five years. Exclusion criteria: Previous or present treatment with immunosuppressive medication or biologicals. Steroid treatment within 30 days of evaluation Evaluation of patients: Baseline brain MRI and PET using 11C-PK11195 and 11C-TMSX with a protocol used in our previous studies. MS functional composite (MSFC), brain atrophy, quantitative diffusion tensor magnetic resonance imaging (DTI-MRI) measures, and neuropsychological status. At 5 years PET using 11C-UCB-J radioligand.

Positron emission tomography (PET) imaging methods: 1) Detection of microglial activation. The investigators shall use the TSPO-ligand 11C-PK11195 to evaluate the level of microglial activation in the NAWM, in normal appearing gray matter (NAGM) and in the periplaque areas. The 11C-PK11195 imaging. 2) A2A-AR detection. The investigators shall investigate the distribution of the A2A-ARs using PET and (11C-TMSX). This will be performed to correlate A2A-AR expression with microglial activation in the central nervous system (CNS) of RRMS patients at risk of converting to SPMS. The 11C-TMSX imaging.3) Evaluation of synaptic density using 11C-UCB-J-PET. The association between 11C-UCB-J binding and cognitive functions will be evaluated.

Based on earlier experience with PET ligands it is estimated that 15 subjects per group is enough to reveal 15% difference in 11C-PK11195 and 11C-TMSX uptake between the study groups with 90% power at p-level <0.05. The correlation analyses between the variables will be performed with Spearman's non-parametric test for non-linear, and Pearson's test for linear association.

Facilities: Turku PET Centre (TPC) is the national PET Centre in Finland. It has six state-of the-art PET scanners and a long history of performing PET scanning in neurological disorders, and in animal models thereof (www.turkupetcentre.fi). Radiochemical synthesis of 11C-PK11195 has been established in TPC and study projects on MS patients have been completed and published by our research group previously. The 11C-TMSX and 11C-UCB-J are already in use in the TPC.

People involved: Dr. Laura Airas, MD, PhD. Consultant in neurology, and assistant professor in neurology. Professor Juha Rinne, MD, Consultant in Neurology. Turku PET Centre. Professor Riitta Parkkola, MD, Neuroradiologist. Dr. Eero Rissanen MD, PhD. Dr. Marcus Sucksdorff, MD, PhD student.

ELIGIBILITY:
Inclusion Criteria:

* RRMS, age 40-50 years, MS-diagnosis for a minimum of five years.

Exclusion Criteria:

* Previous or present treatment with immunosuppressive medication or biologicals. - Steroid treatment within 30 days of evaluation

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Relapsing remitting MS (RRMS) patients on the verge of secondary progression, age 40-50 years, MS-diagnosis for a minimum of five years before entering the study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-04; Primary Completion 2023-12 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of microglial activation and MS progression | 5 years
  11C-PK11195-radioligand binding using PET

SECONDARY OUTCOMES:
Correlation of 11C-TMSX radioligand binding and MS progression | 5 years
  11C-TMSX-radioligand binding using PET
Correlation of 11C-UCB-J-radioligand binding and cognition | 5 years
  Correlation 11C-UCB-J-radioligand binding and cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Laura Airas, MD, Docent, Principal Investigator — Turku University Hospital, division of clinical neurosciences
Locations (1):
- Turku PET Centre, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: Undecided
Multi-center collaboration under discussion

REFERENCES:
- [Derived] Laaksonen S, Sucksdorff M, Vuorimaa A, Kuhle J, Nylund M, Rajander J, Wahlroos S, Matilainen M, Saraste M, Airas L. Predictors of risk of secondary progression in multiple sclerosis. Ther Adv Neurol Disord. 2025 Sep 9;18:17562864251357276. doi: 10.1177/17562864251357276. eCollection 2025. PMID 40951543
- [Derived] Sjoros T, Saraste M, Matilainen M, Nylund M, Koivumaki M, Kuhle J, Leppert D, Airas L. Serum glial fibrillary acid protein associates with TSPO-expressing lesions in multiple sclerosis brain. Ther Adv Neurol Disord. 2025 Jul 28;18:17562864251352998. doi: 10.1177/17562864251352998. eCollection 2025. PMID 40756531